CLINICAL TRIAL: NCT02532712
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Escalation, Phase I Clinical Trial to Evaluate the Safety, Tolerability and PK of EC-18 After Oral Administration in Healthy Male Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and PK of EC-18 After Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC-18-101
Record Dates: First submitted 2015-08-04; First posted 2015-08-26 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Chemotherapy-Induced Neutropenia
Keywords: EC-18; Hematology; Cancer; Neutropenia
MeSH Terms: conditions — Neoplasms; Neutropenia | interventions — 1-palmitoyl-2-linoleoyl-3-acetyl-rac glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- Single dose group-Group 1-Experimental (Experimental): Single dose, 500mg of Study drug(EC-18)
  Interventions: Drug: EC-18
- Single dose group-Group 1-Placebo (Placebo Comparator): Single dose, 500mg of Placebo
  Interventions: Drug: Placebo
- Single dose group-Group 2-Experimental (Experimental): Single dose, 1000mg of Study drug(EC-18)
  Interventions: Drug: EC-18
- Single dose group-Group 2-Placebo (Placebo Comparator): Single dose, 1000mg of Placebo
  Interventions: Drug: Placebo
- Single dose group-Group 3-Experimental (Experimental): Single dose, 2000mg of Study drug (EC-18)
  Interventions: Drug: EC-18
- Single dose group-Group 3-Placebo (Placebo Comparator): Single dose, 2000mg of Placebo
  Interventions: Drug: Placebo
- Single dose group-Group 4-Experimental (Experimental): Single dose, 4000mg of Study drug (EC-18)
  Interventions: Drug: EC-18
- Single dose group-Group 4-Placebo (Placebo Comparator): Single dose, 4000mg of Placebo
  Interventions: Drug: Placebo
- Multiple dose group-Group 1-Experimental (Experimental): Multiple dose, Study drug(EC-18) 500mg, Once daily, for 14 days
  Interventions: Drug: EC-18
- Multiple dose group-Group 1-Placebo (Placebo Comparator): Multiple dose, Placebo 500mg, Once daily, for 14 days
  Interventions: Drug: Placebo
- Multiple dose group-Group 2-Experimental (Experimental): Multiple dose, Study drug(EC-18) 1000mg, Once daily, for 14 days
  Interventions: Drug: EC-18
- Multiple dose group-Group 2-Placebo (Placebo Comparator): Multiple dose, Placebo 1000mg, Once daily, for 14 days
  Interventions: Drug: Placebo
- Multiple dose group-Group 3-Experimental (Experimental): Multiple dose, Study drug(EC-18) 2000mg, Once daily, for 14 days
  Interventions: Drug: EC-18
- Multiple dose group-Group 3-Placebo (Placebo Comparator): Multiple dose, Placebo 2000mg, Once daily, for 14 days
  Interventions: Drug: Placebo
- Multiple dose group-Group 4-Experimental (Experimental): Multiple dose, Study drug(EC-18) 4000mg, Once daily, for 14 days
  Interventions: Drug: EC-18
- Multiple dose group-Group 4-Placebo (Placebo Comparator): Multiple dose, Placebo 4000mg, Once daily, for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EC-18 — EC-18 Soft-capsule (500mg/1 capsule)
  Other Names: EC18 Soft-capsule
  Arms: Multiple dose group-Group 1-Experimental; Multiple dose group-Group 2-Experimental; Multiple dose group-Group 3-Experimental; Multiple dose group-Group 4-Experimental; Single dose group-Group 1-Experimental; Single dose group-Group 2-Experimental; Single dose group-Group 3-Experimental; Single dose group-Group 4-Experimental
Drug: Placebo — Placebo with same shape and size
  Other Names: Placebo for EC-18 (Sofe-capsule)
  Arms: Multiple dose group-Group 1-Placebo; Multiple dose group-Group 2-Placebo; Multiple dose group-Group 3-Placebo; Multiple dose group-Group 4-Placebo; Single dose group-Group 1-Placebo; Single dose group-Group 2-Placebo; Single dose group-Group 3-Placebo; Single dose group-Group 4-Placebo

SUMMARY:
This study is a Dose block-randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Escalation, Phase I clinical trial to assess the safety, tolerability and pharmacokinetics of single-dose and multiple-dose oral administration of the investigational product, EC-18 (study drug) in healthy adult male volunteers.

DETAILED DESCRIPTION:
In vitro and in vivo efficacy studies and clinical trials have shown that EC-18 has a mode of action of improving neutropenia by promoting neutrophil production from hematopoietic stem cells and at the same time, efficiently controlling STAT6/Complement 3(C3), suggesting its potential to be developed as an orally administered new drug for treatment of neutropenia resulting from decreased neutrophils caused by administration of an anticancer agent.

This study is a Dose block-randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Escalation, Phase I clinical trial to assess the safety, tolerability and pharmacokinetics of single-dose and multiple-dose oral administration of the investigational product, EC-18 (study drug) in healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male aged between 19 and 45 years, inclusive, at the time of providing the informed consent form
* Body weight ≥ 50 kg, and calculated BMI in the range of 18.5 kg/m2 ≤ BMI < 25.0 kg/m2 ☞ BMI(body mass index) = Body weight (kg)/[height (m)]2
* No inherited or chronic disease and pathologic symptoms or findings from internal examinations
* Eligible subject based on findings from clinical laboratory tests, such as hematology, blood chemistry, urinalysis and immunoserology, and ECG, as conducted by a responsible doctor depending on characteristics of the drug
* Written consent on voluntary decision of participation and compliance with precautions after being fully informed of and completely understanding this trial
* Consent to practice medically acceptable contraception during the trial

Exclusion Criteria:

* Hypersensitivity to a drug containing an ingredient of the investigational product (EC-18) or similar ingredient (e.g., deer antler) or other drugs (e.g., aspirin, antibiotics) or medical history of clinically significant hypersensitivity
* Active infection such as chronic or local infection based on screening tests or inquiry, verifiable medical records
* Serious infection that required hospitalization or use of antibiotics within 30 days prior to the first dose of the investigational product, based on an inquiry or verifiable medical records
* Presence of a clinically significant hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, nervous, blood, cardiovascular, urogenital, psychiatric disorder or its prior history
* (1) Presenting tuberculosis or prior history of tuberculosis or (2) positive results from a QuantiFERON® -TB Gold in Tube Assay conducted due to a contact with a tuberculosis patient within the past 3 months or signs and symptoms of suspected tuberculosis
* Prior history of a gastrointestinal disorder (e.g., Crohn's disease, ulcer) or surgery (except for simple appendectomy or hernia surgery) that may affect drug absorption, etc.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
No. and severity of Adverse event as a Measure of Safety and Tolerability | From date of D-1 until Follow-up visit: up to 30 days
Vital signs, physical examination, clinical laboratory tests, ECG as a Measure of Safety and Tolerability | From date of screening until Follow-up visit: up to 60 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters of EC-18 following single oral dose: Cmax (Maximum observed plasma drug concentration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following single oral dose: Tmax (Time of maximum drug concentration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following single oral dose: AUClast (Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following single oral dose: AUCinf (Area under the plasma concentration-time curve from time zero extrapolated to the infinite time) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following single oral dose: t1/2 (Half-life) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following single oral dose: CL/F (Apparent total clearance of the drug from plasma after oral administration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Cmax,ss (Maximum (peak) steady-state plasma drug concentration during a dosage interval) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Cmin,ss (Minimum steady-state plasma drug concentration during a dosage interval) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Cavg,ss (Average steady-state plasma drug concentration during multiple-dose administration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Fluctuation | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: t1/2 (half-life) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: AUCτ (Area under the plasma concentration-time curve from time zero to time t) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: AUCinf (Area under the plasma concentration-time curve from time zero to infinity) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Cmax (Maximum (peak) plasma drug concentration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Tmax (Time to reach maximum (peak) plasma concentration following drug | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: CL/F (Apparent total clearance of the drug from plasma after oral administration) | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose
Pharmacokinetic parameters of EC-18 following multiple oral doses: Accumulation index | [0], 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 16, 24, 36, 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Min-Soo Park, Professor, Principal Investigator — Yonsei University Health System, Severance Hospital (Seoul)
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
I will update the status when it is decided.